CLINICAL TRIAL: NCT00175526
Title: PIERS (Pre-eclampsia Integrated Estimate of RiSk) Model: Predicting Adverse Maternal Outcomes in Pre-eclampsia
Brief Title: Predicting Complications in Women With Toxaemia
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H03-70137
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Toxemia
MeSH Terms: conditions — Toxemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: preeclampsia — This research project, 'a severity score for pre-eclampsia,' will develop such a clinical tool that is specific to the condition. To develop and validate the tool w

SUMMARY:
At present, the management of pre-eclampsia is guided by expert opinions that are not well-based on firm evidence. What is required is a clinical tool that can accurately determine a women's risk for adverse outcomes, and thereby reduce the risk for women while safely prolonging pregnancies remote from term (to improve fetal outcomes). This research project, 'a severity score for pre-eclampsia,' will develop such a clinical tool that is specific to the condition. This severity score will be used clinically (to guide management) and in research (in both clinical trials and basic science research), and will provide an evidence base on which to build future practice, improving outcomes for pregnant women and their babies. In addition, this project is part of a three part strategy to better understand the mechanisms of disease in pre-eclampsia and to investigate a potential disease-modifying therapy, namely, recombinant human activated protein C.

DETAILED DESCRIPTION:
In North America, pre-eclampsia ('toxaemia of pregnancy') is the most common cause for women to die during or shortly after pregnancy. It is also the most common reason for babies who are otherwise doing well to be delivered prematurely; this is with the intent purpose of protecting maternal health and safety. In many ways it is similar to the systemic inflammatory response syndrome ('septicaemia').

This project is part of a three part strategy to better understand the mechanisms of disease in pre-eclampsia and to investigate a potential disease-modifying therapy, namely, recombinant human activated protein C. We have surveyed Canadian practice, and undertaken both feasibility and pilot studies for this project.

At present, the management of pre-eclampsia is guided by expert opinions that are not well-based on firm evidence. What is required is a clinical tool that can accurately determine a women's risk for adverse outcomes, and thereby reduce the risk for women while safely prolonging pregnancies remote from term (to improve fetal outcomes). This research project, 'a severity score for pre-eclampsia,' will develop such a clinical tool that is specific to the condition. To develop and validate the tool we will recruit 3000 women in Canada, the UK, and Australasia who are admitted to a hospital with either pre-eclampsia or one of its variants. At the same time, because the majority of deaths associated with pre-eclampsia occur in low and middle income countries, we will recruit 3000 women from Uganda, China, Fiji, South Africa and Pakistan with pre-eclampsia. We will use this cohort to test the model and ensure it accurately predicts risk in this new population.

This severity score will be used clinically (to guide management) and in research (in both clinical trials and basic science research), and will provide an evidence base on which to build future practice, improving outcomes for pregnant women and their babies.

ELIGIBILITY:
Inclusion Criteria:

These criteria reflect the evidence that pre-eclampsia is more than hypertension and proteinuria, particularly at onset:

* Hypertension. sBP >140mmHg and/or dBP >90mmHg, twice, >4h apart after 20 weeks' gestation. sBP will be included to reflect international guidelines.
* Proteinuria. 24h urinary protein >0.3g/d3, or in the absence of a 24h urine collection: >2+ dipstick proteinuria after 20wk or a random protein:creatinine ratio >30mg protein/mmol creatinine106-108.
* HELLP syndrome that is non-hypertensive and non-proteinuric, using Sibai's criteria109,
* One eclamptic seizure without preceding hypertension or proteinuria ('BEST' definition of eclampsia38).
* Women admitted with suspected 'superimposed pre-eclampsia' will also be included (e.g., those with a history of pre-existing hypertension with new proteinuria (>2+) or accelerated hypertension3;23;24).

Exclusion Criteria:

* Occurrence of the maternal outcome (e.g., recurrent eclampsia) prior to collection of the predictors.
* Admission to hospital in spontaneous labour (as clinicians will not attempt to stop these labours).

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women with pre-eclampsia ('toxaemia of pregnancy') which is the most common cause for women to die during or shortly after pregnancy.
Sampling Method: Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2005-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To identify the maternal and fetal variables predictive of a combined adverse maternal outcome occurring within one week of hospital admission for pre-eclampsia | Unknown at this time

SECONDARY OUTCOMES:
To identify whether these also predict the combined adverse maternal outcome at any time following admission ii to identify whether these variables can predict a combined adverse perinatal outcome both (a) within one week and (b) at any time foll | Unknown at this time

CONTACTS AND LOCATIONS:
Overall Officials: Peter von Dadelszen, MD, Principal Investigator — University of British Columbia
Locations (6):
- Canada (4):
  - Children's and Women's Health Centre of BC, Vancouver, British Columbia
  - Kingston General Hospital, Kingston, Ontario
  - Ottawa Hospital-General Campus, Ottawa, Ontario
  - le Centre hospitalier universitaire de Sherbrooke, Sherbrook, Quebec
- Christchurch Women's Hospital, Christchurch, New Zealand
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom